CLINICAL TRIAL: NCT05052203
Title: Researching the Effects of Sepsis on Quality Of Life, Vitality, Epigenome and Gene Expression During RecoverY From Sepsis (REQOVERY)
Brief Title: Researching the Effects of Sepsis on Quality Of Life, Vitality, Epigenome and Gene Expression During RecoverY From Sepsis
Acronym: REQOVERY
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Hjalmar Bouma (Other)
Responsible Party: Sponsor-Investigator, Hjalmar Bouma, Internist and Research Fellow, University Medical Center Groningen
Organization: University Medical Center Groningen (Other)
Other Study IDs: 202100108
Record Dates: First submitted 2021-08-27; First posted 2021-09-22 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Sepsis; Infection
Keywords: Post sepsis syndrome; Epigenetic; Transcriptome; Recovery
MeSH Terms: conditions — Sepsis; Infections | interventions — Epigenesis, Genetic; Gene Expression; Gene Expression Profiling; Leukocyte Count

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Exposure of interest: study DNA methylation (epigenetics) and gene expression (transcriptomics) of blood leukocytes — The primary objective is to study DNA methylation (epigenetics) and gene expression (transcriptomics) of blood leukocytes between sepsis survivors at ED admission and three months after hospital discharge

SUMMARY:
Sepsis is a life-threatening dysregulated immune response to infection associated with multi-organ failure and a high mortality rate.While researchers have focused mainly on acute sepsis, post-sepsis care of survivors has long been neglected despite the observation that many sepsis survivors suffer from debilitating post-sepsis syndrome. This syndrome is characterized by frequent hospital readmissions and increased mortality due to persistent immune dysfunction, cardiovascular disease, and cognitive impairment, causing poor quality of life and a substantial burden on the healthcare system. Disconcertingly, the number of sepsis survivors at risk for hospital readmission continues to rise.7 Of the post-sepsis symptoms, post-sepsis immunosuppression is perhaps the most clinically important. While sepsis presents as an initial phase of hyperinflammation (a "cytokine storm"), it is followed by an immunosuppressive phase that is now understood to last weeks to months and predisposes survivors to lethal secondary infections and sepsis recurrence. A third of deaths eight years post-sepsis are caused by recurrent sepsis.We hypothesize that changes in the transcriptome and DNA methylome in immune cells of survivors might be the underlying driver for prolonged immunosuppression, and may also be correlated with long-term morbidity and mortality post-sepsis, as well as other symptoms of post-sepsis syndrome including PTSD and cardiovascular disease.

ELIGIBILITY:
Inclusion criteria sepsis group:

* Adult patients, aged between 18 and 85 years
* Able to provide informed consent themselves or informed consent can be obtained via next of kin or legal guardian
* Included in Acutelines, where blood sample was drawn upon ED admission
* Satisfy the Sepsis-3 criteria for sepsis (Figure 2), combined with clinical suspicion of infection and/or fever (body temperature > 38.5°C)
* Survive at 3 months post discharge
* Inclusion criteria control group:Adult patients, aged between 18 and 85 years
* Able to provide informed consent themselves or informed consent can be obtained via next of kin or legal guardian
* Included in Acutelines, where blood sample was drawn upon ED admission
* Non-infectious reason of admission (specifically syncope, electrolyte disturbance, intoxication, gastro-intestinal bleeding)

4.3 Exclusion criteria

The participants should not meet any of the following exclusion criteria:

* Transfer from another hospital
* Emergency room visit in connection with accidental exposure of bodily material to patient ("needle stick injury")
* Visit an emergency room in connection with organ transplantation
* Discharged home without hospital admittance after ED visit
* Unable to give blood
* Immunosuppressive therapies such as corticosteroids (>10mg) or small molecule immune suppressants within the last three months, or biologicals administered within the last year
* Radiotherapy or systemic chemotherapy within the last three months
* Known pregnancy; the presence of pregnancy will be verified by asking the potential participant
* A hospitalization of more than 21 days

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients between 18-85 years old admitted to the emergency department (ED) of the University Medical Center Groningen (UMCG) with suspected sepsis according to the sepsis-3 criteria who survive their ED admission at three months. A control group will compose of age and sex-matched ED patients admitted for non-infectious causes. Both the septic patients and controls have already been enrolled in the Acutelines study.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-09-28 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
DNA methylation (epigenetics) using the Illumina MethylationEPIC kit. Changes in DNA methylation at gene promoter/enhancer sites will be correlated through the NetworkAnalyst platform. | baseline versus 3 months follow up
  The primary objective of the current project is to measure changes in DNA methylation (i.e. epigenetics) of blood leukocytes between sepsis survivors at ED admission and three months after hospital discharge.
Gene expression (transcriptomics/qPCR) will be measured using the Illumina Hi-Seq instrument. Differential gene expression will be correlated through the NetworkAnalyst platform. | baseline versus 3 months follow up
  The primary objective of the current project is to measure changes in gene expression (i.e. transcriptomics) of blood leukocytes between sepsis survivors at ED admission and three months after hospital discharge.

SECONDARY OUTCOMES:
Nutrition status measured with PS-SGA Short Form and SNAQ form. (both questionnaires) | 3 months
  study the association between epigenetic and transcriptomic signatures in sepsis and survivors with nutrition status. PS-SGA short form looks at weight loss, upper arm circumference, apetite and functionallity. PS-SGA short form scores weight, food intake, symptoms, activities and functionalilyti (nummeric; 0-52).
Mortality. Mortality status will be obtained from the Municipal Personal Records Database (BRP), containing reliable and complete registration all Dutch citizens | 1 year
  study the association between epigenetic and transcriptomic signatures and mortality in sepsis survivors and non-survivors and healthy controls. Mortality will be retrieved from the electronic health records (EHR) from the hospital and municipal registration. The cause of death will be retrieved from the EHR from the hospital, general practitioner and Dutch statistics' office (CBS).
Demographics | 3 months
  To study the association between epigenetic and transcriptomic signatures in sepsis survivors with demographics. Information about demograpics will be retrieved from the electronic health records (EHR) from the hospital.
Intoxications | 3 months
  To study the association between epigenetic and transcriptomic signatures in sepsis survivors with intoxications. Information about intoxications will be retrieved from the electronic health records (EHR) from the hospital.
Medication use | 3 months
  To study the association between epigenetic and transcriptomic signatures in sepsis survivors with medication use. Medication use will be retrieved from the electronic health records (EHR) from the hospital, general practitioner and pharmacy.
Sepsis severity defined with SOFA score | 3 months follow up
  study the association between severity of sepsis and the epigenetic and transcriptomic signatures in sepsis. SOFA scores will be available for patients admitted because of an infection.
Fatigue assessed with piper fatigue scale | 3 months
  To study the association between epigenetic and transcriptomic signatures in sepsis and survivors with fatigue.Piper Fatigue Scale-12 (PFS-12; 0-10, higher scores reflect more fatigue among four subscales (a) behavior, (b) affect, (c) sensory, (d) cognition)
Mood assessed with the Patient Health Questionnaire-2 ( (questionnaire) | 3 months
  To study the association between epigenetic and transcriptomic signatures in sepsis and survivors with mood. Patient Health Questionnaire-2 (PHQ-2; 0-6, higher score corresponds to reduced mental health)
Somatic symptoms (e.g. Patient Health questionnaire-15) | 3 months
  To study the association between epigenetic and transcriptomic signatures in sepsis and survivors with somatic symptoms. Patient Health Questionnaire-15 (PHQ-15; 0-30, minimal-high somatic symptom severity)
Activities of daily living as determined by EQ-5D-5L (if abnormal also Katz-ADL-6) | 3 months
  To study the association between epigenetic and transcriptomic signatures in sepsis and survivors with activities of daily living. EuroQol-5D (EQ5D; simple descriptive profile and a single index value for health status; higher values corresponding with better health) with visual analogue scale (VAS; 0-100, worse-best experienced health). Katz ADL-6 (0-6, fully dependent-independent)
Physical activity (e.g. Short Questionnaire to Assess Health-Enhancing Activity) (SQUASH) and 'Utrechtse activiteiten lijst' (UAL)) | 3 months
  To study the association between epigenetic and transcriptomic signatures in sepsis and survivors with physical activity
Co-morbidity (a.o. Charlson comorbidity index) | 3 months
  To study the association between epigenetic and transcriptomic signatures in sepsis and survivors with comorbidity. Co-morbidity will be retrieved from the electronic health records (EHR) from the hospital, general practitioner and pharmacy. Data will be registered according to the Charlson' co-morbidity index (CCI; 1-2 mild co-morbidity, 3-4 moderate co-morbidity, 5 severe co-morbidity)
Vital parameters | At baseline and three months.
  Heart rate (bpm), blood pressure (mmHg), oxygen saturation (SpO2, SaO2, PaO2), breathing frequency (per min), consciousness (Glasgow coma scale), pain score (VAS), nausea/vomiting (y/n), defecation (y/n), urination (y/n), body weight (kg), length (cm), fluid balance (ml/day).
Length-of-stay in hospital/intensive care unit (ICU) | 0-3 months
  Length-of-stay in hospital and on intensive care unit (ICU) in days

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No